CLINICAL TRIAL: NCT01328093
Title: A Phase 3, Multicenter, Double-Blind Comparison of LY2140023 and Aripiprazole in Patients With DSM-IV-TR Schizophrenia Followed by Open-Label Treatment With LY2140023
Brief Title: A Comparison Study of LY2140023 and Aripiprazole in Schizophrenia Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision to stop the trial was based on efficacy results in the overall schizophrenia participant population.
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14211; H8Y-MC-HBDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2140023 (Experimental): Double Blind Phase: 40 milligrams (mg) administered orally, given twice daily for 24 weeks. Dose may be adjusted to a minimum of 20 mg or a maximum of 80 mg. Open Label Phase: 40 mg administered orally, given twice daily for an additional 28 weeks.
  Interventions: Drug: LY2140023
- Aripiprazole (Active Comparator): Double Blind Phase: 15 mg administered orally, given once daily for 24 weeks. Dose can be adjusted to a minimum of 10 mg or a maximum of 30 mg. Open Label Phase: LY2140023, 40 mg administered orally, given twice daily for an additional 28 weeks.
  Interventions: Drug: LY2140023; Drug: Aripiprazole

INTERVENTIONS:
Drug: LY2140023 — Administered orally
Drug: Aripiprazole — Administered orally
  Arms: Aripiprazole

SUMMARY:
The purpose of this study is to determine whether weight gain will be significantly less in LY2140023 than aripiprazole in patients with schizophrenia.

DETAILED DESCRIPTION:
The primary objective of this study was to test the hypothesis that mean weight gain, as assessed by change from baseline, would be statistically significantly less for flexibly dosed LY2140023 (20, 40, or 80 mg twice daily [BID]) than for flexibly dosed aripiprazole (10, 15, or 30 mg/day) in patients with schizophrenia after 24 weeks of double-blind treatment.

This was a multicenter, randomized, double-blind, Phase 3 study to assess the safety and efficacy of LY2140023 (flexibly dosed between 20 and 80 mg BID) in patients with schizophrenia. An active control, aripiprazole (flexibly dosed between 10 and 30 mg/day), was included for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Female participants of childbearing age must test negative for pregnancy at screening and agree to use single, effective, medically acceptable method of birth control
* Participants must require initiation of or modification to current antipsychotic treatment as outpatients
* Participants must be considered reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and be willing to perform all study procedures
* Participants must be able to understand the nature of the study and have given their own informed consent

Exclusion Criteria:

* Have been on treatment with aripiprazole in the past 2 months or are aripiprazole nonresponders
* Participants who are pregnant, nursing, or intend to become pregnant within 30 days of completing the study
* Hospitalized within 2 weeks of screening or have been hospitalized for an exacerbation of symptoms of schizophrenia with a discharge date in the past 2 months
* Participants who are actively suicidal
* Participants with uncorrected narrow-angle glaucoma, history of or current seizure disorder, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, uncontrolled thyroid condition or other serious or unstable illnesses
* Participants who have had electroconvulsive therapy (ECT) within 3 months prior to screening or will have ECT at any time during the study
* Participants with known medical history of Human Immunodeficiency Virus positive (HIV+) status
* Test positive for (1) Hepatitis C virus antibody or (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody
* Participants with a corrected QT interval (Bazett's; QTcB)>450 milliseconds (msec) (male) or >470 msec (female) at screening
* Participants who have a history of inadequate clinical response to antipsychotic treatment for schizophrenia
* Participants who have received treatment with any depot formulation of an antipsychotic medication within 1 dosing interval, minimum of 4 weeks, prior to screening
* Are currently enrolled in, or discontinued within the last 60 days from, a clinical trial involving an investigational product or unapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have any other psychiatric diagnoses in addition to schizophrenia
* Have previously completed or withdrawn from this study, or any other study investigating LY2140023 or any predecessor molecules with glutamatergic activity
* Participants who have received an adequate treatment trial, in the opinion of the investigator, with clozapine at doses greater than 200 milligrams (mg) daily within 12 months prior to screening, or who have received any clozapine at all during the month before screening
* Diagnosis of substance-induced psychosis within 7 days of screening (or at any time during the study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (32):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cerritos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Gables, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sanford, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Creve Coeur, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Princeton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willingboro, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresh Meadows, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeSoto, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wharton, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottignies
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulon
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oranienburg
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vic
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luleå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo

REFERENCES:
- [Derived] Adams DH, Zhang L, Millen BA, Kinon BJ, Gomez JC. Pomaglumetad Methionil (LY2140023 Monohydrate) and Aripiprazole in Patients with Schizophrenia: A Phase 3, Multicenter, Double-Blind Comparison. Schizophr Res Treatment. 2014;2014:758212. doi: 10.1155/2014/758212. Epub 2014 Mar 19. PMID 24772351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 24-week Double-Blind Active Treatment Phase and was followed by a 28-week Open-Label Active Treatment Phase. Modified intent-to-treat (mITT) is all randomized participants who received at least 1 dose of study drug, excluding participants from a Good Clinical Practice (GCP) noncompliant study site.
Groups:
- LY2140023-DB / LY2140023-OL: 40 milligrams (mg) LY2140023 administered orally, twice daily for 24 weeks during the Double-Blind (DB) Phase. Dose was adjustable to 20 mg twice daily or 80 mg twice daily.
  40mg LY2140023 administered orally, twice daily for 28 weeks during the Open -Label (OL) Phase. Dose was adjustable to 20 mg twice daily or 80 mg twice daily.
- Aripiprazole-DB / LY2140023-OL: 15 mg aripiprazole administered orally, once daily for 24 weeks during the Double-Blind (DB) Phase. Dose was adjustable to 10 mg once daily or 30 mg once daily.
  40mg LY2140023 administered orally, twice daily for 28 weeks during the Open -Label (OL) Phase. Dose was adjustable to 20 mg twice daily or 80 mg twice daily.
Period: Double-Blind Phase
Arm/Group | LY2140023-DB / LY2140023-OL | Aripiprazole-DB / LY2140023-OL
Started | 516 | 162
Received at Least 1 Dose of Study Drug | 514 | 161
Modified Intent-To-Treat (mITT) | 511 | 161
Completed | 231 (Not all participants entered Open-Label Treatment Phase.) | 84 (Not all participants entered Open-Label Treatment Phase.)
Not Completed | 285 | 78
Not completed — Adverse Event | 78 | 15
Not completed — Withdrawal by Subject | 42 | 14
Not completed — Lost to Follow-up | 39 | 14
Not completed — Protocol Violation | 30 | 10
Not completed — Lack of Efficacy | 55 | 13
Not completed — Sponsor Decision | 17 | 3
Not completed — Entry Criteria Not Met | 7 | 5
Not completed — Scheduling conflict | 8 | 3
Not completed — Subject is moving or has moved | 8 | 1
Not completed — Death | 1 | 0
Period: Open-Label Phase
Arm/Group | LY2140023-DB / LY2140023-OL | Aripiprazole-DB / LY2140023-OL
Started | 200 | 73
Received at Least 1 Dose of Study Drug | 198 | 73
Modified Intent-To-Treat (mITT) | 197 | 73
Completed | 60 | 23
Not Completed | 140 | 50
Not completed — Sponsor Decision | 98 | 34
Not completed — Protocol Violation | 8 | 3
Not completed — Lost to Follow-up | 10 | 1
Not completed — Adverse Event | 10 | 4
Not completed — Lack of Efficacy | 5 | 6
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Scheduling conflict | 2 | 1
Not completed — Subject is moving or has moved | 2 | 0
Not completed — Entry Criteria Not Met | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) population: All randomized participants who received at least 1 dose of study drug, excluding participants from the excluded study site.
Groups:
- LY2140023-DB: 40 milligrams (mg) LY2140023 administered orally, twice daily for 24 weeks during the Double-Blind (DB) Phase. Dose was adjustable to 20 mg twice daily or 80 mg twice daily.
- Aripiprazole-DB: 15 mg aripiprazole administered orally, once daily for 24 weeks during the Double-Blind (DB) Phase. Dose was adjustable to 10 mg once daily or 30 mg once daily.
- Total: Total of all reporting groups
Arm/Group | LY2140023-DB | Aripiprazole-DB | Total
Number analyzed (Participants) | 511 | 161 | 672
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.29 (10.86) | 42.95 (10.95) | 42.45 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 55 | 240
  Male | 326 | 106 | 432
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 23 | 96
  Not Hispanic or Latino | 438 | 138 | 576
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 6
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 238 | 64 | 302
  White | 259 | 93 | 352
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 21 | 6 | 27
  United States | 341 | 112 | 453
  Puerto Rico | 27 | 6 | 33
  Spain | 19 | 6 | 25
  Belgium | 13 | 3 | 16
  Poland | 20 | 7 | 27
  Romania | 21 | 6 | 27
  Austria | 6 | 2 | 8
  Germany | 26 | 9 | 35
  Sweden | 17 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks in Body Weight
Description: Mixed model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigator, visit, prior olanzapine use, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had baseline and at least one post-baseline weight measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 487 | 155
kilograms (kg) | -2.8 (0.4) | 0.4 (0.6)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p < 0.001, Type III Tests — No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = -3.2, Standard Error of Mean 0.7

2. Secondary Outcome: Percentage of Participants With Clinically Significant Weight Change
Description: Clinically significant change in body weight is defined as either an increase or decrease in weight of ≥7% from baseline.
Time Frame: Baseline up to 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline weight measurement, excluding participants from the excluded study site.
Measure: Number; unit: percentage of participants
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 488 | 155
percentage of participants
  ≥7% Increase | 4.1 | 7.1
  ≥7% Decrease | 13.1 | 3.2
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.110, Cochran-Mantel-Haenszel — P-value is for ≥7% increase
Statistical Analysis 2: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is for ≥7% decrease

3. Secondary Outcome: Change From Baseline up to 24 Weeks in Barnes Akathisia Scale (BAS)
Description: The BAS is a 4-item instrument that evaluates akathisia associated with use of antipsychotic medications. Item 4 Global Clinical Assessment of Akathisia is rated on a 6- point scale, with scores range from 0 (no symptoms) to 5 (increased severity of symptoms); Only Item 4 was analyzed and presented. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline BAS global score measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 455 | 141
units on a scale | 0.00 (0.03) | -0.04 (0.04)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.353, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 0.04, Standard Error of Mean 0.04

4. Secondary Outcome: Change From Baseline up to 24 Weeks in Simpson-Angus Scale (SAS)
Description: The SAS is used to measure Parkinsonian-type symptoms in participants exposed to antipsychotics. SAS consists of 10 items, each rated on a 5-point scale: 0 (complete absence of the condition) to 4 (presence of the condition in extreme form). The SAS Total Score is obtained by adding the ten items, and ranges from 0 to 40. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment by-visit-interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline SAS total score measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 456 | 141
units on a scale | -0.17 (0.06) | -0.20 (0.08)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.698, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 0.03, Standard Error of Mean 0.09

5. Secondary Outcome: Change From Baseline up to 24 Weeks in Abnormal Involuntary Movement Scale (AIMS)
Description: AIMS is a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 to 10 are rated on a 5- point scale: 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Items 11 and 12 are yes/no questions regarding the dental condition of a participant. The AIMS 1-7 Total Score is the sum of Items 1 through 7 of the AIMS, and ranges from 0 to 28. Higher scores indicate greater severity of illness. Only AIMS 1-7 Total Score was analyzed and presented. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline AIMS 1-7 Total Score measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 456 | 141
units on a scale | -0.11 (0.05) | -0.10 (0.07)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.924, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = -0.01, Standard Error of Mean 0.07

6. Secondary Outcome: Change From Baseline up to 24 Weeks in Positive and Negative Syndrome Scale (PANSS) Total and Subscale Scores
Description: The PANSS consists of 30 items and 3 subscales and is designed to measure severity of psychopathology in schizophrenia. The PANSS Positive Subscale and the PANSS Negative Subscale each contain 7 items, and the remaining 16 items make up the PANSS General Psychopathology Subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). The PANSS Total Score is the sum of the 30 items, with scores range from 30 to 210. The PANSS Positive Subscale and PANSS Negative Subscale scores each range from 7 to 49. The PANSS General Psychopathology subscale score ranges from 16 to 112. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline PANSS measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 482 | 155
units on a scale
  PANSS Total Score | -12.03 (0.99) | -15.58 (1.58)
  PANSS Positive Score: number analyzed (Participants) | 482 | 154
  PANSS Positive Score | -3.40 (0.32) | -4.62 (0.50)
  PANSS Negative Score | -2.98 (0.31) | -3.34 (0.48)
  PANSS General Psychopathology Score | -5.80 (0.56) | -7.85 (0.89)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.045, Type III Tests — P-value is for PANSS Total Score. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = 3.55, Standard Error of Mean 1.77
Statistical Analysis 2: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.032, Type III Tests — P-value is for PANSS Positive Score. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = 1.21, Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.509, Type III Tests — P-value is for PANSS Negative Score. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = 0.36, Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.040, Type III Tests — P-value is for PANSS General Psychopathology Score. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = 2.05, Standard Error of Mean 1.00

7. Secondary Outcome: Change From Baseline up to 24 Weeks in EuroQol-5 Dimensions Questionnaire (EQ-5D) Visual Analog Scale (VAS) Health State Score
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument that contains 2 parts: a health status profile and a visual analog scale (VAS) to rate global health-related quality of life. VAS health state scores range from 0 (worst imaginable health state) to 100 (best imaginable health state). The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline VAS health state measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 386 | 126
units on a scale | 4.2 (1.4) | 3.1 (2.0)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.601, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 1.1, Standard Error of Mean 2.1

8. Secondary Outcome: Schizophrenia Resource Utilization Module (S-RUM) - Number of Emergency Room (ER) or Equivalent Facility Visits and Outpatient Medical Visits
Description: The S-RUM is a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, ER visits, and outpatient medical visits for a specified period of time. Item 1 asks about the number of ER or equivalent facility visits a participant had for psychiatric (psych) illness. Item 2 asks about the number of ER or equivalent facility visits a participant had for non-psychiatric (non-psych) illness or injury. Item 5 asks about the number of outpatient visits to other physicians (not psychiatrists or dentists). Analysis of variance (ANOVA) was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for pooled investigator, gender and treatment.
Time Frame: Baseline to 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug and had S-RUM assessment, excluding participants from the excluded study site. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: visits
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 451 | 146
visits
  ER/Facility (Psych) visits | 0.06 (0.01) | 0.04 (0.02)
  ER/Facility (Non-Psych) visits | 0.06 (0.01) | 0.02 (0.02)
  Outpatient (Non-Psych or Dentist) visits | 0.28 (0.04) | 0.30 (0.06)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.322, Type III Tests — P-value is for ER/Facility (Psych) visits. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = -0.02, Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.099, Type III Tests — P-value is for ER/Facility (Non-Psych) visits. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = -0.04, Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.787, Type III Tests — P-value is for Outpatient (Non-Psych or Dentist) visits. No adjustments for multiple comparisons were made. The treatment comparison was evaluated at a 2-sided significance level of 0.05; LS Mean Differences = 0.02, Standard Error of Mean 0.07

9. Secondary Outcome: Schizophrenia Resource Use Module (S-RUM) - Number of Sessions With a Psychiatrist
Description: The S-RUM is a 31-item questionnaire to assess the participant's occupation (work and home), living arrangements, encounters with law enforcement, victimization, emergency room (ER) visits, and outpatient medical visits for a specified period of time. Item 4 asks about the number of sessions with a psychiatrist a participant had. Analysis of variance (ANOVA) was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for pooled investigator, gender and treatment.
Time Frame: Baseline to 24 weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: sessions
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 451 | 146
sessions | 0.39 (0.07) | 0.41 (0.11)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.892, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 0.02, Standard Error of Mean 0.12

10. Secondary Outcome: Change From Baseline up to 24 Weeks in Subjective Well-Being Under Neuroleptic Treatment Scale- Short Form (SWN-SF) Total Score
Description: The SWN-SF measures subjective well-being of the participant for the previous 7 days. The 20-item scale covers 5 health domains (subscales; 4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). Each of the 5 subscale scores range from 4 to 24. SWN-SF Total Scores range from 20 to 120. Higher scores indicate greater well-being. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline SWN-SF Total Score measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 423 | 133
units on a scale | 4.6 (1.0) | 5.3 (1.5)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.630, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = -0.8, Standard Error of Mean 1.6

11. Secondary Outcome: Change From Baseline up to 24 Weeks in Personal and Social Performance (PSP) Score
Description: The PSP scale is a 100-point (minimum 1, maximum 100), single item, clinician-rated scale to assess a participant's overall functioning, including personal and social relationships, socially useful activities, self-care, and disturbing and aggressive behaviors. Higher scores indicate a higher level of functioning. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline PSP measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 431 | 136
units on a scale | 5.9 (0.7) | 6.4 (1.1)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.679, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = -0.5, Standard Error of Mean 1.2

12. Secondary Outcome: Change From Baseline up to 24 Weeks in Clinical Global Impression-Severity Scale (CGI-S)
Description: The CGI-S instrument is used to record the severity of mental illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline CGI-S measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 487 | 155
units on a scale | -0.51 (0.05) | -0.69 (0.08)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.055, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 0.17, Standard Error of Mean 0.09

13. Secondary Outcome: Change From Baseline up to 24 Weeks in 16-Item Negative Symptom Assessment (NSA-16)
Description: The NSA-16 scale is used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale rates participants on 16 "anchors". Each item ("anchor") is rated from 1 (better) to 6 (worse). The NSA-16 Total Score is the sum of the 16 specific items and ranges from 16 to 96. Higher scores indicate greater severity of illness. The Mixed Model Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and standard error. LS mean values were adjusted for baseline, treatment, gender, pooled investigative site, visit, predefined subpopulation, treatment-by-visit interaction and baseline-by-visit interaction.
Time Frame: Baseline, 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline NSA-16 Total Score measurement, excluding participants from the excluded study site.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 431 | 136
units on a scale | -6.22 (0.68) | -6.37 (1.03)
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.891, Type III Tests — [p-value comment as in outcome 1, analysis 1]; LS Mean Differences = 0.15, Standard Error of Mean 1.11

14. Secondary Outcome: Number of Participants With 30% or Greater Decrease in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (absence of symptoms) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS Total Score and ranges from 30 to 210. Higher scores indicate greater severity of illness. Data presented are the number of participants with 30% or greater decrease from baseline in PANSS Total score.
Time Frame: Baseline up to 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline PANSS measurement, excluding participants from the excluded study site. Last observation carried forward (LOCF) principle was used.
Measure: Number; unit: participants
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 486 | 155
participants | 133 | 49

15. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Measured by Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Data presented are the number of participants with treatment-emergent suicidal ideation or behavior during the treatment period (with a change from lead-in baseline in C-SSRS).
Time Frame: Baseline to 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline C-SSRS measurement, excluding participants from the excluded study site.
Measure: Number; unit: participants
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 488 | 155
participants
  Treatment-Emergent Suicidal Ideation | 46 | 7
  Treatment-Emergent Suicidal Behavior | 7 | 0
Statistical Analysis 1: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.064, Fisher Exact — P-value is for Treatment-Emergent Suicidal Ideation
Statistical Analysis 2: Comparison: LY2140023-DB vs Aripiprazole-DB; Test type: Superiority or Other; p = 0.205, Fisher Exact — P-value is for Treatment-Emergent Suicidal Behavior

16. Secondary Outcome: Time to Discontinuation
Description: The time to discontinuation due to any reason was defined as the total number of days between randomization and discontinuation date. The time to discontinuation was analyzed using Kaplan-Meier estimated survival curves. Participants who completed the study were considered censored.
Time Frame: Randomization up to 24 weeks
Population: Modified intent-to-treat (mITT) population: All randomized participants who received at least one dose of study drug, excluding participants from the excluded study site. Participants who completed the study were considered censored: 229 for LY2140023 group and 84 for Aripiprazole group.
Measure: Median (Full Range); unit: days
Arm/Group | LY2140023-DB | Aripiprazole-DB
Number analyzed (Participants) | 511 | 161
days | 140 [120 to 158] | 169 [131 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Description: Adverse events were reported for all randomized participants who received at least 1 dose of study drug, excluding participants from a Good Clinical Practice (GCP) noncompliant study site.
Groups:
- LY2140023-OL: 40mg LY2140023 administered orally, twice daily for 28 weeks during the Open -Label (OL) Phase, following the treatment with either 40 mg LY2140023 or 15 mg aripiprazole during the Double-Blind Phase. Dose was adjustable to 20 mg twice daily or 80 mg twice daily.
Arm/Group | LY2140023-DB | Aripiprazole-DB | LY2140023-OL
Serious Adverse Events (participants affected / at risk) | 42/511 | 5/161 | 12/270
Other Adverse Events (participants affected / at risk) | 358/511 | 107/161 | 112/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2140023-DB (N=511) | Aripiprazole-DB (N=161) | LY2140023-OL (N=270)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1/185 (1) | 0/55 (0) | 0/106 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Event was determined not to be a seizure by Seizure Adjudication Committee.
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Event resulted in death.
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 8 (8) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 15 (16) | 2 (2) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2140023-DB (N=511) | Aripiprazole-DB (N=161) | LY2140023-OL (N=270)
Left atrial dilatation (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 13 (14) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (15) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 20 (21) | 8 (9) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 99 (112) | 18 (19) | 15 (15)
Toothache (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 41 (58) | 12 (14) | 5 (8)
Fatigue (General disorders) | 14 (14) | 6 (6) | 0 (0)
Irritability (General disorders) | 11 (11) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (5) | 1 (1)
Therapeutic response unexpected (General disorders) | 6 (6) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 38 (40) | 8 (10) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 2 (2) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 2/185 (2) | 0/55 (0) | 1/106 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 29 (30) | 4 (4) | 3 (3)
Weight decreased (Investigations) | 9 (9) | 1 (1) | 2 (2)
Weight increased (Investigations) | 9 (9) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22) | 6 (6) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 9 (9) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (6) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (2) | 3 (3)
Akathisia (Nervous system disorders) | 13 (13) | 12 (12) | 2 (2)
Disturbance in attention (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 16 (16) | 8 (9) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 57 (69) | 10 (10) | 16 (17)
Myoclonus (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1)
Sedation (Nervous system disorders) | 4 (4) | 4 (4) | 2 (2)
Somnolence (Nervous system disorders) | 15 (17) | 4 (5) | 2 (2)
Tremor (Nervous system disorders) | 8 (10) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 21 (22) | 8 (8) | 6 (8)
Bruxism (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 4 (4) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 50 (53) | 19 (20) | 8 (9)
Restlessness (Psychiatric disorders) | 9 (10) | 2 (2) | 1 (1)
Schizophrenia (Psychiatric disorders) | 11 (12) | 0 (0) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1/326 (1) | 2/106 (2) | 0/164 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0/185 (0) | 1/55 (1) | 0/106 (0)
Female sterilisation (Surgical and medical procedures) | 0/185 (0) | 1/55 (1) | 0/106 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early. 97% of participants had completed or discontinued from the DB Phase prior to termination. Outcome measure populations excluded data from a site that had significant GCP noncompliance issues (3 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days